CLINICAL TRIAL: NCT05991310
Title: Evaluating the Safety and Efficacy of Telemedicine Neurology Assessments on a Mobile Stroke Unit
Acronym: MSU-TELEMED
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Melbourne Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023.110
Record Dates: First submitted 2023-07-27; First posted 2023-08-14 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Ischemic Stroke; Intracerebral Hemorrhage
Keywords: mobile stroke unit; stroke
MeSH Terms: conditions — Ischemic Stroke; Cerebral Hemorrhage; Stroke

STUDY DESIGN:
Intervention Model Description: The days in which the neurologist will be on or off the mobile stroke unit will be randomly determined. Randomization will be stratified by nurse category (Nurse Practitioner versus Clinical Nurse Consultant) with an adaptive component to balance the number of patients reviewed in person or via telemedicine within each nurse category. The randomized schedule will be generated in a rolling fashion on a weekly basis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telemedicine Assessment by Remote Neurologist (Experimental): Following the initial assessment, the stroke nurse will activate the telemedicine video conference call and review the patient with the telemedicine neurologist. The telemedicine neurologist will perform a NIHSS with assistance from the stroke nurse, and this will be documented on the clinical records. Imaging will be evaluated remotely by the telemedicine neurologist. If there is a decision to administer thrombolysis, the stroke neurologist and nurse will discuss treatment with the patient or next of kin, where appropriate and able, to acquire assent in a timely manner.
  Interventions: Other: Telemedicine Assessment by Remote Neurologist
- In-Person Assessment by an Onboard Neurologist (Active Comparator): Upon arrival on-scene, the MSU stroke nurse, neurologist, and paramedic will liaise with local ambulance services to obtain initial clinical details and perform an initial assessment. The NIHSS will be performed by the neurologist, and this will be documented on standardized clinical records. Imaging will be assessed at the console available within the ambulance. If there is a decision to administer thrombolysis, the stroke neurologist and nurse will discuss treatment with the patient or next of kin, where appropriate and able, to acquire assent in a timely manner.
  Interventions: Other: In-Person Assessment by an Onboard Neurologist

INTERVENTIONS:
Other: Telemedicine Assessment by Remote Neurologist — Use of a telemedicine platform for a neurologist, remotely located, to assess a MSU patient, review imaging, and decide on the required treatments.
  Arms: Telemedicine Assessment by Remote Neurologist
Other: In-Person Assessment by an Onboard Neurologist — Traditional in-person assessment of a patient by a neurologist located onboard the MSU
  Arms: In-Person Assessment by an Onboard Neurologist

SUMMARY:
The goal of this clinical trial is to compare a telemedicine neurologist staffing model to a traditional on-board model in patients being assessed for suspected acute stroke on a mobile stroke unit.

DETAILED DESCRIPTION:
This study is a prospective randomized mobile stroke unit trial comparing two staffing models: 1) a neurologist reviewing the patient via telemedicine (intervention) versus 2) an onboard neurologist assessing the patient in-person (comparator). Daily periods of remote (telemedicine) or in person (onboard) neurologist assessments will be randomly determined using an adaptive design.

ELIGIBILITY:
Inclusion Criteria:

1. Adults >=18 years of age
2. Presenting within 24 hours of symptom onset or last known well.
3. Patients assessed by MSU without cancellation (either by the local ambulance team or by MSU) prior to attending the patient.

Exclusion Criteria:

1. Attendance of the Melbourne MSU is deemed unnecessary by either the local paramedic team or the MSU team based on provided information prior to arrival on scene.
2. The patient presents significant medical or logistical challenges which greatly delay standard treatment.
3. Any other medical contraindication at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Desirability of Outcome Ranking (DOOR) of: Safety, Scene-to-decision Treatment Times, and Resource Efficiency | See pre-specified outcome section for details
  The odds that a random participant treated through a telemedicine assessment will have a more desirable DOOR scale outcome than a random participant treated by an onboard neurologist. Such a odds is referred to as the Win Ratio, as it reflects the odds of a random participant treated via telemedicine "winning" against a random participant treated via an onboard model in a direct one-to-one comparison.
  The design evaluates, in order of importance: Safety, Scene-to-decision time metrics, Resource efficiency
  If a participant in one treatment arm is achieving better safety than the comparator, this is defined as a "win" for that participant and a "loss" for the comparator. If there is no difference in safety, time to treatment decision is compared. If no clinically meaningful difference is observed, then resource utilization is compared. If there is no difference in resource utilization, the two participants are declared as tied for the overall outcome.

SECONDARY OUTCOMES:
On-scene to eyes-on-patient (for the neurologist) | Time of Acute Assessment on the Mobile Stroke Unit (up to 2 hours from arrival on scene)
On-scene to imaging | Time of Acute Assessment on the Mobile Stroke Unit (up to 2 hours from arrival on scene)
On-scene to imaging review by the neurologist | Time of Acute Assessment on the Mobile Stroke Unit (up to 2 hours from arrival on scene)
On-scene to definitive decision making | Time of Acute Assessment on the Mobile Stroke Unit (up to 2 hours from arrival on scene)
  Inclusive of the following: 1) Decision for thrombolysis, 2) Decision to refer for endovascular thrombectomy, 3) Decision to stand down case, or 4) Decision to transfer to stroke hospital (e.g. suspected stroke but unable to treat on MSU)
90-Day mRS | 90 days (+/- 10 days from symptom onset)
  Clinical outcomes for patients who receive thrombolysis on the MSU or are transferred to a comprehensive center for endovascular clot retrieval

OTHER OUTCOMES:
Safety Outcomes | Up to 72 hours from symptom onset
  1. Clinician unable to complete assessment
  2. Post-thrombolysis Complications
  3. Deterioration during assessment
Scene-to-decision Treatment Times | Up to 2 hours from arrival on-scene
Resource Efficiency | Up to 12 hours (duration of MSU working hours)
  Evaluated as the proportion of productive time the neurologist is actively involved in the care of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Vignan Yogendrakumar, MD PhD, Principal Investigator — Melbourne Health; Anna H Balabanski, MD PhD, Principal Investigator — Melbourne Health
Locations (1):
- Royal Melbourne Hospital Mobile Stroke Unit, Melbourne, Victoria, Australia

REFERENCES:
- [Background] Yogendrakumar V, Balabanski AH, Johns H, Churilov L, Parsons NK, Beharry J, Weir L, Yassi N, Zhao H, Warwick A, Coote S, Langenberg F, Branagan L, Siddiqi W, Bivard A, Campbell BCV, Donnan GA, Davis SM; MSU-TELEMED Investigators dagger. Evaluating the Safety and Efficacy of Telemedicine Physician Assessments on a Mobile Stroke Unit: Protocol for a Prospective Open-Label Blinded End-Point Randomized Controlled Trial. J Am Heart Assoc. 2024 Nov 5;13(21):e036856. doi: 10.1161/JAHA.124.036856. Epub 2024 Oct 18. PMID 39424402
- [Derived] Yogendrakumar V, Balabanski AH, Johns H, Churilov L, Mutimer CA, Barker J, Parsons NK, Shin SJ, Beharry J, Weir L, Yassi N, Zhao H, Warwick A, Coote S, Langenberg F, Branagan L, Siddiqi W, Hocking G, Ng FC, Sanders LM, Choi PMC, Wijeratne T, Crompton DE, Ma H, Cloud G, Campbell BCV, Donnan GA, Davis SM. A Randomized Trial of Telemedicine Models of Care on a Mobile Stroke Unit. NEJM Evid. 2025 Dec 22:EVIDoa2500217. doi: 10.1056/EVIDoa2500217. Online ahead of print. PMID 41429047
- See also: Statistical Analysis Plan — https://www.medrxiv.org/content/10.1101/2025.02.11.25322103v1